CLINICAL TRIAL: NCT02923206
Title: Proof-of-Concept Trial on Selective Removal of the Antiangiogenic Factor Soluble Fms-like Tyrosine Kinase-1 (sFlt-1) in Pregnant Women With Preeclampsia Via Apheresis Utilizing the Flt-1 Adsorption Column
Brief Title: Proof-of-Concept Trial on Selective Removal of sFlt-1 in Pregnant Women With Preeclampsia Via Apheresis
Acronym: SAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2016-313
Record Dates: First submitted 2016-09-19; First posted 2016-10-04 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Preeclampsia
Keywords: apheresis; pregnancy; pre-eclampsia; PE; sFlt-1; Pre-term
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 0 - healthy volunteers (Experimental): Phase 0 is an initial safety phase where subjects will undergo one single TheraSorb sFlt-1 adsorber apheresis procedure.
  Interventions: Device: TheraSorb sFlt-1 adsorber
- Phase A - preeclampsia patients (Experimental): Phase A is a safety and dose-finding phase during which pregnant women diagnosed with preeclampsia will undergo one single TheraSorb sFlt-1 adsorber apheresis procedure.
  Interventions: Device: TheraSorb sFlt-1 adsorber
- Phase B - preeclampsia patients (Experimental): Phase B is a safety and efficacy phase during which pregnant women diagnosed with preeclampsia will undergo TheraSorb sFlt-1 adsorber apheresis procedures up to twice weekly.
  Interventions: Device: TheraSorb sFlt-1 adsorber

INTERVENTIONS:
Device: TheraSorb sFlt-1 adsorber — Removal of excessive sFlt-1 from the plasma of subjects/ patients with therapeutic apheresis.

SUMMARY:
This clinical investigation is a medical device trial to examine the safety and efficacy of TheraSorb sFlt-1 adsorber treatment of pregnant patients with preeclampsia.

ELIGIBILITY:
Reduced criteria!

Phase 0

Inclusion Criteria:

* Age ≥18 and ≤45 years;
* Male or female;
* Female subjects of childbearing potential must have a negative serum pregnancy test result at screening and practice two reliable methods of contraception throughout the study.

Exclusion Criteria:

* Dysfunction of cerebral nervous system and/or heart disease;
* History of preexisting chronic renal disease;
* Treatment with ACE inhibitors;
* Therapeutic full anticoagulation therapy prior to trial entry;
* Liver abnormalities;
* Clinically significant pulmonary edema and/or thrombocytopenia and/or anemia;
* Active hepatitis B, C, or tuberculosis infection or HIV infection
* Hypersensitivity to heparin and/or citrate;
* Indications that prohibit transient anticoagulation using heparin and/or ACD-A-solutions;
* Known intolerance to extracorporeal procedures in general or towards one of the individual excipients or towards other supporting agents;
* Drug or alcohol abuse within the last 2 years;
* Lack of compliance of subject;
* History or diagnosis of severe periodontitis;

Phase A and B

Inclusion Criteria:

* Age >18 and ≤45 years ;
* Pregnant woman with pre-term preeclampsia
* sFlt-1/PlGF ratio ≥85 ;
* sFlt-1 level of ≥ 8000pg/mL

Exclusion Criteria:

Maternal exclusion criteria

* History of cardiac impairments including uncontrolled arrhythmia, unstable angina, decompensated congestive heart failure or valve disease;
* History of preexisting chronic renal disease (CKD stage >3a, eGFR ≤45ml/min/1.73m²);
* Treatment with ACE inhibitors;
* Therapeutic full anticoagulation therapy prior to trial entry;
* Signs or history of clinically significant cerebral nervous system dysfunction;
* History of clinically significant liver abnormalities;
* Clinically significant pulmonary edema and/or thrombocytopenia and/or anemia;
* Active hepatitis B, C, tuberculosis infection or HIV-positive status;
* Any condition that the investigator deems a risk to the patient or fetus in completing the trial;
* Indications that prohibit transient anticoagulation using heparin and/or ACD-A-solutions;
* Drug or alcohol abuse within the last 2 years;
* Lack of compliance of patient;
* Known intolerance to extracorporeal procedures in general or to one of the excipients or other supporting agents;
* Hypersensitivity to heparin and/or citrate;
* < 30 0/7 weeks of gestation and abnormal CTG and/or abnormal Ductus venosus Doppler flow,
* ≥30 0/7 weeks of gestation and Doppler evidence of umbilical artery Absent or Reversed End-Diastolic Velocity (AREDV);
* Various Placental exclusion criteria;
* Multiple pregnancy
* History or diagnosis of severe periodontitis

Fetal exclusion criteria

* Any known trisomy;
* Amniotic fluid index <5cm (greatest single pocket <2cm);
* Estimated fetal weight <3rd percentile for gestational age;
* Fetus which are at high risk of heart disease;
* Fetus with congenital heart defect;
* Fetal signs of bleeding;
* Hydrops fetalis;
* Pathological fetal Doppler flow of the ductus venosus (absent A-wave in two measurements);
* Evidence of severe fetal malformations;
* Known infection of fetus;
* Known severe anemia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of AEs and SAEs in healthy volunteers until the 2 weeks follow-up (Phase 0) | until 2 weeks post treatment
Occurrence of AEs and SAEs in pregnant subjects and the fetus or infant until the 6 weeks post-delivery visit is reached (Phase A-B). | until 6 weeks post delivery

SECONDARY OUTCOMES:
Phase 0: Determine changes of sFlt-1 levels. | until 2 weeks post treatment
Phase 0: Complement activation levels pre-, during and post apheresis. | Before, during and directly following the performance of the single apheresis treatment (1 day)
Phase 0: Concentration of antibody leaching during an apheresis procedure | During an apheresis procedure (1 day)
Phase 0: Change of HAMA levels in pre- and post apheresis blood | until 2 weeks post treatment
Phase 0: Evaluate blood pressure values | until 2 weeks post treatment
Phase 0: Evaluate spot urine values | until 2 weeks post treatment
Phase A/B: Occurrence of SAEs in the one year follow-up period | until end of FU, (1 year)
Phases A/B: Evaluate antibody leaching in phase A. | During the performance of the single apheresis treatment in Phase A (1 day) as well as pre and 3hrs post apheresis
Phases A and B: Evaluate maternal sFlt-1 levels. | Constant measures throughout the trial until delivery (up to 19 weeks)
Phases A/B: Evaluate the sFlt-1/PlGF ratio. | Constant measures throughout the trial until delivery (up to 19 weeks)
Phases A/B:Evaluate neonatal umbilical cord blood sFlt-1 levels at birth. | at birth
Phases A/B: Determine HAMA levels | until 6 week FU visit
Phases A/B: Time and method of delivery, and anesthesia administered | at birth
Phases A and B: Determine the post-partum maternal and neonatal length of hospitalization. | Following birth up to one year
Phases A/B: Evaluate standard markers of fetal development throughout pregnancy. | From start of trial until delivery (up to 19 weeks)
Phases A/B: Evaluate standard markers of neonatal development. | Directly following delivery until end of FU (1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Benzing, Prof. Dr., Principal Investigator — University Clinic Cologne
Locations (4):
- Germany (2):
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Leipzig, Leipzig
- United Kingdom (2):
  - Cambridge Clinical Trials Unit, Addenbrooke's Hospital, Cambridge
  - Oxford University Hospitals NHS Foundation Trust, John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No